CLINICAL TRIAL: NCT04995549
Title: Construction of a Mechanical Data Base for Mathematically Modeling Uncertainties in Human Skin Tissues
Brief Title: SKin Uncertainties Modeling
Acronym: SKUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/527
Record Dates: First submitted 2021-05-19; First posted 2021-08-09 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Unrecognized Condition
Keywords: skin, non lesional, arm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measures using Cutiscan® CS 100 (Experimental)
  Interventions: Device: Cutiscan® CS 100

INTERVENTIONS:
Device: Cutiscan® CS 100 — Repeated measures on healthy volunteers skin (forearm) are performed using Cutiscan® CS 100 device

SUMMARY:
The study is based on measurement device and will provide a database of viscoelastic properties of the forearm skin among healthy volunteers.

These data will be used to develop a mathematical model representative of the mechanical behavior of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 50 years old
* non-opposition to participating in SKUM study
* Affiliation to french social security

Exclusion Criteria:

* Refusal to participate
* Volunteer with any skin disease likely to interfere with the primary outcome
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and / or weak cooperation
* Subject without health insurance
* Pregnant woman
* Subject being in the period of exclusion from another study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Height of displacement (mm) of a skin disc. | Month 1
  The displacement will be obtained from repeated measures, on 30 volunteers, on forearm skin, and using Cutiscan® CS100 device. A database of skin viscoelasticity measure will be built from such data.

CONTACTS AND LOCATIONS:
Overall Officials: Brice CHATELAIN, MD, Principal Investigator — CHU DE BESANCON
Locations (1):
- CHU de besançon, Besançon, France